CLINICAL TRIAL: NCT01792544
Title: Clinical Reminders in Test Reports to Improve Guideline Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Heidenreich, Staff Physician, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SUIRB-021780
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Echocardiography

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statement (Experimental): A statement is added to the echocardiography report describing if and when a follow-up echocardiogram is recommended. The statement may be positive (e.g. follow-up recommended in 6 months) or negative (e.g. no follow-up recommended).
  Interventions: Other: Statement
- No Statement (Experimental): No statement is added to the echocardiography report
  Interventions: Other: No Statement

INTERVENTIONS:
Other: Statement
  Arms: Statement
Other: No Statement
  Arms: No Statement

SUMMARY:
This study examines the impact of adding a statement to the echocardiography report that advises anyone reading the report regarding if and when a follow-up study is recommended.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing echocardiography where the physician creating the report feels a comment is appropriate regarding when follow-up should or should not occur.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1706 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Inappropriate follow-up | 1 year
  Performance of a follow-up echocardiogram when it was not indicated or not performing for a follow-up echocardiogram when it was indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto HCS, Palo Alto, California, United States